CLINICAL TRIAL: NCT07058519
Title: The Efficacy and Safety of Osimertinib-based Adaptive Treatment Guided by Circulating Tumour DNA (ctDNA) Epidermal Growth Factor Receptor Mutation-positive (EGFRm) Dynamic Monitoring in Locally Advanced or Metastatic EGFRm Non-small Cell Lung Cancer (NSCLC) Participants With ctDNA EGFRm Clearance After First-line Osimertinib Plus Chemotherapy: A Phase II, Multicentre, Prospective Study (Adaptive)
Brief Title: A Study of Osimertinib-based Adaptive Treatment Guided by ctDNA EGFRm+ Monitoring in NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Lu Shun, Professor Chief of Shanghai Lung Cancer Center, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-24-22779
Record Dates: First submitted 2025-06-16; First posted 2025-07-10 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic EGFRm Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; EGFRm+; Osimertinib
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (EGFRm ctDNA Clearance Group) (Experimental): EGFRm ctDNA Clearance Group
  Interventions: Drug: Osimertinib-based adaptive treatment
- Cohort 2 (ctDNA EGFRm non-clearance group) (Experimental)
  Interventions: Drug: Osimertinib 80 MG

INTERVENTIONS:
Drug: Osimertinib-based adaptive treatment — Participants in Cohort 1 will receive Osimertinib-based adaptive treatment (either Osimertinib monotherapy or Osimertinib plus chemotherapy) depending on ctDNA EGFRm clearance or relapse by ctDNA EGFRm dynamic monitoring, until radiological disease progression (PD) as per RECIST v1.1 or other withdrawal criteria are met.
  Arms: Cohort 1 (EGFRm ctDNA Clearance Group)
Drug: Osimertinib 80 MG — Participants in Cohort 2 will receive Osimertinib 80 mg once daily (QD) plus pemetrexed maintenance every 3 weeks (Q3W) until radiological PD as per RECIST v1.1 or other withdrawal criteria are met.
  Arms: Cohort 2 (ctDNA EGFRm non-clearance group)

SUMMARY:
The goal of this adaptive, interventional study is to assess the efficacy and safety of osimertinib-based adaptive treatment based on ctDNA dynamic monitoring in locally advanced or metastatic EGFRm NSCLC participants with ctDNA EGFRm clearance after osimertinib plus chemotherapy. The main questions it aims to answer are: 1) PFS during adaptive treatment period in Cohort 1 defined as from initiation of Osimertinib in adaptive period to progression per investigator assessment; 2) Time from initiation of osimertinib in adaptive period to first ctDNA EGFRm relapse or death

DETAILED DESCRIPTION:
Locally advanced or metastatic EGFR mutation-positive (EGFRm) non-small cell lung cancer (NSCLC) (Stage IIIB, IIIC, IV, or recurrent) has a poor prognosis. The 5-year survival rate for metastatic disease is only 8.9%.

While combination therapy with osimertinib and platinum-pemetrexed chemotherapy, as validated by the FLAURA2 trial, has demonstrated improved progression-free survival (PFS), it also introduces increased toxicity, treatment burden, and reduced quality of life. Notably, a subset of patients-approximately 25-30%-achieves long-term benefit from osimertinib monotherapy alone, highlighting the potential to personalize treatment intensity.

Emerging evidence supports circulating tumor DNA (ctDNA) as a dynamic biomarker for guiding therapy. Analyses from FLAURA2 and other studies have shown that early ctDNA EGFRm clearance strongly correlates with superior PFS and can identify patients who may not require continuous combination therapy. Adaptive strategies based on ctDNA clearance have enabled treatment de-escalation in early-stage and advanced NSCLC settings, maintaining efficacy while reducing toxicity. This trial builds on that rationale, aiming to validate ctDNA-guided adaptive therapy to balance efficacy, safety, and quality of life in EGFRm NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent form (ICF) prior to any study specific procedures.
2. Male or female participants aged 18 years old and above.
3. ECOG PS of 0-1.
4. Life expectancy of at least 3 months at recruitment.
5. Participants able to collect plasma samples at baseline.
6. Newly diagnosed, and histologically documented locally advanced or metastatic non-squamous NSCLC with sensitizing EGFR mutations positive (either Exon 19 deletion or 21 L858R, confirmed by histology or cytology), and classified as stage IIIB, IIIC, IV or recurrent NSCLC which are not amenable to curative surgery or radiotherapy (per Version 8 of the International Association for the Study of Lung Cancer [IASLC] Staging Manual in Thoracic Oncology).
7. Detectable EGFRm (Ex19del or L858R) in plasma ctDNA by central Super ARMS PCR testing at the time of screening.
8. Participants must have untreated advanced NSCLC and intend to receive osimertinib plus chemotherapy as first-line treatment. Prior adjuvant and neo-adjuvant therapies (chemotherapy, radiotherapy, immunotherapy, biologic therapy, investigational agents), or definitive radiation/chemoradiation with or without regimens including immunotherapy, biologic therapy, investigational agents, are permitted as long as treatment was completed at least 12 months prior to receiving the first dose of study treatment.
9. Participants with asymptomatic and stable central nervous system (CNS) metastases for at least 2 weeks (for those who received definitive therapy and steroids, a stable neurological status for at least 2 weeks after completion of the treatment is required) will be allowed, including leptomeningeal metastases.
10. At least 1 lesion, not previously irradiated that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have a short axis of ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI), and that is suitable for accurate repeated measurements. If only 1 measurable lesion exists, it is acceptable to be used (as a target lesion) as long as it has not been previously irradiated and as long as it has not been biopsied within 14 days of the baseline tumour assessment scans.
11. Patients with hepatitis B virus (HBV) are only eligible for inclusion if they meet all the following criteria:

    * Demonstrated absence of hepatitis C virus (HCV) co-infection or history of HCV co-infection
    * Demonstrated absence of human immunodeficiency virus (HIV) infection
    * Participants with active HBV infection are eligible if they are:

      * Receiving anti-viral treatment for at least 6 weeks prior to study treatment, HBV DNA is suppressed to <100 IU/mL and transaminase levels are below upper limit of normal (ULN).
    * Participants with a resolved or chronic HBV infection are eligible if they are:

      * Negative for hepatitis B surface antigen (HBsAg) and positive for hepatitis B core antibody [anti-HBc IgG or total anti-HBc Ab]. In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment.

    or
    * Positive for HBsAg, but for > 6 months have had transaminases levels below ULN and HBV DNA levels below <100 IU/mL or below the detectable limit of locally available test kit (i.e., are in an inactive carrier state). In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment.
12. Patients with HIV are only eligible for inclusion if they meet all the following criteria:

    * Demonstrated absence of HBV/ HCV co-infection
    * Undetectable viral RNA load for 6 months
    * CD4+ count of >350 cells/μL
    * No history of AIDS-defining opportunistic infection within the past 12 months
    * Stable for at least 4 weeks on the same anti-HIV medications
13. Females must be using highly effective contraceptive measures, and must have a negative pregnancy test prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal defined as aged 50 years or more and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.
    * Women under 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution.
    * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
14. Male participants must be willing to use barrier contraception.

Exclusion Criteria:

1. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
2. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the participant to participate in the trial or which would jeopardize compliance with the protocol, or active infection (e.g. participants receiving treatment for infection) including hepatitis C and HIV, or active uncontrolled HBV infection. Screening for chronic conditions is not required.
3. Any of the following cardiac criteria:

   * Mean resting corrected QTc >470 msec, obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value.
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g., complete left bundle branch block, third degree heart block and second degree heart block.
   * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as electrolyte abnormalities including:

     * Serum/plasma magnesium* < LLN
     * Serum/plasma calcium* < LLN
     * Hypokalaemia* ≥ CTCAE Grade 2 heart failure, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes.

       * Correction of electrolyte abnormalities should be documented prior to first dose
4. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count (ANC) <1.5 × 109/L
   * Platelet count <100 × 109/L
   * Hemoglobin <90 g/L
   * Alanine aminotransferase (ALT) >2.5 times the ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases.
   * Aspartate aminotransferase (AST) >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases.
   * Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
   * Serum Creatinine >1.5 times ULN concurrent with creatinine clearance <50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
5. Any concurrent and/or other active malignancy that has required treatment within 2 years of first dose of investigational product (IP).
6. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2 prior platinum-therapy related neuropathy.
7. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
8. Prior treatment with any systemic anti-cancer therapy for advanced NSCLC not amenable to curative surgery or radiation including chemotherapy, biologic therapy, immunotherapy, or any investigational drug. Prior adjuvant and neo-adjuvant therapies (chemotherapy, radiotherapy, immunotherapy, biologic therapy, investigational agents), or definitive radiation/chemoradiation with or without regimens including immunotherapy, biologic therapies, investigational agents are permitted as long as treatment was completed at least 12 months prior to the development of recurrent disease.
9. Prior treatment with an EGFR-TKI.
10. Major surgery within 4 weeks of the first dose of IP. Procedures such as placement of vascular access, biopsy via mediastinoscopy or biopsy via video assisted thoracoscopic surgery (VATS) are permitted.
11. Palliative radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of IP.
12. Participants currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of cytochrome P450 (CYP) 3A4 (at least 3-week prior). All participants must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
13. Participation in another clinical study with an investigational product within 5 half-lives of the compound or 3 months whichever is greater prior to Day 1.
14. History of hypersensitivity to active or inactive excipients of Osimertinib or drugs with a similar chemical structure or class to Osimertinib.
15. Contraindication for pemetrexed and cisplatin/carboplatin according to local approved label.
16. Women who are breast-feeding.
17. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).
18. Judgment by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2029-01-24 (Estimated); Study Completion 2029-01-24 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) in Cohort 1 | From initiation of osimertinib in the adaptive therapy period until radiological disease progression or death (up to 33 months).
  Progression-Free Survival (PFS) is defined as the time from the first dose of osimertinib during the adaptive treatment period to the first documentation of disease progression based on investigator assessment according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1, or death from any cause, whichever occurs first.
Time to First ctDNA EGFRm Relapse or Death in Cohort 1 | From initiation of osimertinib in the adaptive therapy period until ctDNA EGFR mutation relapse or death (up to 33 months)
  Time to ctDNA EGFR mutation-positive (EGFRm) relapse is defined as the time from the start of osimertinib treatment in the adaptive therapy period to the first detection of EGFRm in plasma circulating tumour DNA (ctDNA), as assessed by Super ARMS PCR, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) in Cohort 1 | From initiation of osimertinib in adaptive therapy period until death (up to 33 months)
  Overall Survival (OS) is defined as the time from the first dose of osimertinib in the adaptive therapy period to death from any cause. The 24-month landmark survival rate will be reported.
Cumulative Duration of Chemotherapy Holiday in Cohort 1 | From start of adaptive therapy to disease progression or death (up to 33 months)
  The cumulative duration (in weeks) that participants in Cohort 1 receive osimertinib monotherapy without chemotherapy will be calculated during the adaptive treatment period.
Progression-Free Survival (PFS) in Cohort 2 | From initiation of maintenance therapy to radiological disease progression or death (up to 33 months)
  PFS in Cohort 2 is defined as the time from the start of osimertinib plus pemetrexed maintenance therapy to the first documentation of disease progression per RECIST v1.1 or death from any cause.
Overall Survival (OS) in Cohort 2 | From initiation of maintenance therapy to death (up to 33 months)
  OS is defined as the time from the first dose of osimertinib plus pemetrexed maintenance therapy to death from any cause. The 24-month landmark survival rate will be reported.
Change from Baseline in Health-Related Quality of Life Scores (EORTC QLQ-C30) | From baseline through end of treatment (up to 33 months)
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) (0-100) will be used to evaluate participants' health-related quality of life. Higher scores on the QLQ-C30 indicate bad life quality of patient. Change from baseline in domain scores will be analyzed. The higher the score is, the worse the quality of life is.
Change from Baseline in Lung Cancer-Specific Symptoms (EORTC QLQ-LC13) | From baseline through end of treatment (up to 33 months)
  The EORTC QLQ-LC13 questionnaire will be used to assess lung cancer-specific symptoms (e.g., cough, dyspnea), with score range 0-100. Higher scores on the QLQ-LC13 indicate worse symptom severity. Changes from baseline will be reported.

OTHER OUTCOMES:
Frequency of ctDNA EGFRm Relapse During Osimertinib Monotherapy in Cohort 1 | From start of osimertinib monotherapy to disease progression or switch to combination therapy (up to 33 months)
  The proportion of participants who experience re-emergence of ctDNA epidermal growth factor receptor mutations (EGFRm) during osimertinib monotherapy in the adaptive therapy period will be reported, as assessed by Super ARMS PCR.
Correlation Between ctDNA EGFRm Relapse and Disease Progression Events | From adaptive therapy initiation to progression (up to 33 months)
  The temporal and statistical correlation between ctDNA EGFRm re-detection and radiological disease progression events will be analyzed.
Acquired Resistance Mechanisms at Disease Progression | At time of disease progression (up to 33 months)
  Acquired resistance mechanisms will be assessed using next-generation sequencing (NGS) of plasma (mandatory) and optional tumor tissue samples collected at the time of disease progression. Alterations may include gene mutations, amplifications, and immune markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No